CLINICAL TRIAL: NCT04349670
Title: Safety and Efficacy of GPOEM in the Treatment of Gastroparesis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pier Alberto Testoni, Professor, IRCCS San Raffaele
Other Study IDs: GPOEM
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Gastroparesis; Gastroparesis Postoperative; Gastroparesis With Diabetes Mellitus
Keywords: GPOEM; gastroparesis; pyloromyotomy
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: GPOEM - gastric per-oral endoscopic myotomy — Endoscopic section of the pyloric muscle with submucosal tunnel technique.

SUMMARY:
The purpose of this study is to assess the clinical efficacy and safety in the treatment of gastroparesis.

DETAILED DESCRIPTION:
After being informed about the data collected, all the patients affected with gastroparesis undergoing Gastric Per-Oral Endoscopic Myotomy (GPOEM) will be included in the observational protocol.

Data concerning pre-operative symptoms and results of the imaging studies will be recorded together with operative time and operative complications.

Patients will undergo periodical clinical consults and gastric emptying scintigraphy to assess the improvement in the symptoms and gastric motility.

ELIGIBILITY:
Inclusion Criteria:

* Gastroparesis (GCSI > 2 OR Gastric emptying half-time > 180 min OR gastric retention at 120 min > 60% OR good response to botulinum if former criteria not met)

Exclusion Criteria:

* Age < 18 years
* Inability to understand protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected with clinical or scintigrafic severe gastroparesis or patients with moderate symptoms/gastric scintigraphic delayed emptying with good response to botulinum.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | 1, 3, 6, 12, 24 months
  Change in symptomatological scores
Functional efficacy | 3, 12, 24 months
  Change of scintigraphy evaluated gastric emptying time
Complications | peri-operative time (48 hours)
  Evaluation of the operative adverse events

SECONDARY OUTCOMES:
Correlation of symptoms | 3, 12, 24 months
  Evaluate the correlation between symptoms and gastric emptying

CONTACTS AND LOCATIONS:
Locations (1):
- Pier Alberto Testoni, Milan, Italy

IPD SHARING:
Plan to Share IPD: No